CLINICAL TRIAL: NCT00406471
Title: Rubeosis Anti-VEGF (RAVE) Trial for Ischemic Central Retinal Vein Occlusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Greater Houston Retina Research (Other)
Responsible Party: Principal Investigator, David M. Brown, M.D., Director of Research, Greater Houston Retina Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAVE; NCT00406471
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Ischemic Central Retinal Vein Occlusion
Keywords: Ischemic; Central; Retinal; Vein; Occlusion; Ranibizumab; Lucentis; CRVO; ISCRVO
MeSH Terms: conditions — Ischemia; Bites and Stings | interventions — Ranibizumab

ARMS (2):
- 1 (Active Comparator): 500 micrograms of ranibizumab
  Interventions: Drug: Ranibizumab (Lucentis)
- 2 (Active Comparator): 300 microgram ranibizumab
  Interventions: Drug: Ranibizumab (Lucentis)

INTERVENTIONS:
Drug: Ranibizumab (Lucentis) — 500 microgram intravitreal injection for 8 months or 300 microgram intravitreal injection for 8 months

SUMMARY:
The RAVE (Rubeosis Anit-VEgf) trial, utilizes monthly intravitreal Ranibizumab (Lucentis) injections for 9 months to see if total VEGF blockade will prevent neovascular glaucoma and eliminate the need for panretinal photocoagulation in patients with ischemic central retinal vein occlusion.

DETAILED DESCRIPTION:
The most devastating complication of ischemic CRVO is the development of anterior segment neovascularization and the resulting morbidity from neovascular glaucoma. This complication appears to be directly correlated with intraocular VEGF levels. Currently there is no proven treatment to decrease the formation of rubeosis. Current management of the disease consists of pan-retinal photocoagulation once significant anterior segment neovascularization becomes manifest. This treatment destroys peripheral retina (with peripheral retinal field) and presumably works by eventually lowering ocular VEGF levels which causes secondary regression of rubeosis.

As ranibizumab blocks VEGF, this treatment when delivered intraocularly may prevent neo-vascular glaucoma while preserving peripheral visual fields in this patient population.

Risks of intravitreal injections are well known and include endophthalmitis and retinal detachment. This risk should be less than 1% with proper injection technique and experienced retinal surgeons. As the incidence of neovascular glaucoma (with resultant loss of central and peripheral visual fields) is approximately 50% in ischemic CRVO, the small risk of intravitreal injection is warranted if the drug shows efficacy. In a small number of subjects in previous animal and human trials, intraocular pressure was acutely elevated when the drug volume was placed intravitreally. An eye with a compromised circulation (such as ischemic CRVO) may experience less perfusion if this occurred. Previous intravitreal studies of ranibizumab have not utilized anterior chamber paracentesis to compensate for the volume of intravitreal drug to be placed. This was reasonable because an eye with a normal retinal circulation can tolerate relatively high intraocular pressure for a limited time. This protocol for this study will include anterior chamber paracentesis prior to intravitreal injection to minimize this potential risk.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Ischemic CRVO within 3 months of enrollment as per the following inclusion criteria
* Three of the following clinical tests must be present to demonstrate ischemic CRVO:

  * VA 20/200 or worse
  * RAPD 0.9 LU or worse
  * Loss of 1-2e isopter on Goldmann Visual field (Kwon et al. 2001)
  * ERG demonstrating b wave amplitude less than 60% of A wave

Exclusion Criteria:

* Angle neovascularization greater than 3 clock hours with IOP over 30 (Neovascular glaucoma)
* Any previous retinal laser photocoagulation to the study eye
* Any previous intravitreal injection in study eye (triamcinolone or other)
* Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery)
* Intracapsular cataract extraction (posterior capsule needs to be present)
* Previous history of retinal detachment in study eye
* Any previous radiation treatments to head/ neck
* Inability to assess iris neovascularization (corneal opacity precluding gonioscopy)
* Significant cardiovascular disease or cancer that would prevent follow-up visits or completion of the 12 month study
* Significant diabetic retinopathy in the fellow eye (diabetic macular edema, proliferative diabetic retinopathy, or high-risk non-proliferative diabetic retinopathy)
* Pregnancy (positive pregnancy test)
* Prior enrollment in any study for vein occlusion in the study eye
* Participation in another simultaneous medical investigator or trial
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., DME AMD, ocular histoplasmosis, or pathologic myopia)
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period
* Aphakia or absence of the posterior capsule in the study eye
* Previous violation of the posterior capsule is also excluded unless it occurred as a result of YAG laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* History of idiopathic or autoimmune uveitis in either eye
* Structural damage to the center of the macula in the study eye preexisting to CRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s)
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
* Ocular inflammation (including trace or above) in the study eye
* Uncontrolled glaucoma (defined as intraocular pressure ≥30 mm Hg despite treatment with anti- medications) or previous filtration surgery in the study eye
* Infectious blepharitis, keratitis, scleritis, or conjunctivitis (in either eye) or current treatment for serious systemic infection
* Spherical equivalent of the refractive error in the study eye of more than -8 diopters myopia (For patients who have had refractive or cataract surgery in the study eye, pre-operative spherical equivalent refractive error of more than -8 diopters myopia is not allowed) Systemic Conditions
* Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period
* Uncontrolled diabetes mellitus
* Renal failure requiring dialysis or renal transplant
* Premenopausal women not using adequate contraception
* Previous participation in other studies of investigational drugs (excluding vitamins and minerals) within 3 months preceding Day 0
* History of other disease, metabolic dysfunction, physical examination finding, or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications
* INR ≥ 3.0 (e.g. due to current treatment with warfarin). The use of aspirin is not an exclusion.

Other

* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow up procedures
* History of allergy to humanized antibodies or any component of the ranibizumab formulation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Preservation of 5Ve isopter Goldmann visual field versus baseline at 1 year | 12 and 24 months
Estimate the % of subjects progressing to neovascular glaucoma requiring pan-retinal photocoagulation or glaucoma surgery after treatment with ranibizumab (comparing 0.3mg to 0.5mg doses) | 12 and 24 mponths

SECONDARY OUTCOMES:
Assess the systemic and local safety of 0.3mg and 0.5mg of ranibizumab in patients with ischemic CRVO | 12 and 24 months
Assess improvement from baseline in Visual Acuity at 1 year | 12 and 24 months
Assess the impact on retinal thickness and volume (as measured by OCT) | 12 and 24 months
Assess the impact of ranibizumab (0.3mg and 0.5mg) on time to improvement in visual acuity | 12 and 24 months
Asses the impact of ranibizumab (0.3mg and 0.5mg) on time to improvement in retinal thickness | 12 and 24 months
Asses the impact of ranibizumab (0.3mg and 0.5mg) on percentage of patients developing 3 or more clock hours of rubeosis at 6 and 12 months and 24 months | 6, 12, and 24 months
Assess the impact of ranibizumab (0.3mg and 0.5mg) on prevention of greater than 3 clock hours rubeosis (as measured by iris fluorescein angiography) | 12 and 24 months
Assess the impact of ranibizumab on the gain or decrease of area of visual field on 14e Goldman visual field area | 12 and 24 months
Assess the impact of ranibizumab on b wave component of ERG | 12 and 24 months
Aqueous VEGF levels | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David M Brown, MD, Principal Investigator — Vitreoretinal Consultants
Locations (1):
- Vitreoretinal Consultants, Houston, Texas, United States

REFERENCES:
- [Derived] Wykoff CC, Brown DM, Croft DE, Major JC Jr, Wong TP. Progressive retinal nonperfusion in ischemic central retinal vein occlusion. Retina. 2015 Jan;35(1):43-7. doi: 10.1097/IAE.0000000000000277. PMID 25102193
- [Derived] Wykoff CC, Brown DM, Croft DE, Wong TP. Two Year SAVE Outcomes: 2.0 mg ranibizumab for recalcitrant neovascular AMD. Ophthalmology. 2013 Sep;120(9):1945-6.e1. doi: 10.1016/j.ophtha.2013.06.030. No abstract available. PMID 24001533
- See also: Related Info — http://www.houstonretina.com